CLINICAL TRIAL: NCT06874998
Title: Effects of "Parenting in Sweden" on Trust in Social Services - a Randomized Controlled Trial
Brief Title: Effects of "Parenting in Sweden" on Trust in Social Services
Acronym: PiSRCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm City Council (Unknown); Children's right in society (Unknown)
Responsible Party: Principal Investigator, David Ebbevi, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-06868-01
Record Dates: First submitted 2025-02-18; First posted 2025-03-13 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Parent-Child Relations; Immigrant
Keywords: Parental support programs; Parenting; Immigrant parents; Trust in social services; Cultural adaptation

STUDY DESIGN:
Intervention Model Description: Parenting in Sweden (Pis) will be evaluated in a prospective, multicenter, RCT in a ratio of 1:1 to be block randomized to intervention or control group. The groups will be given the same questionnaires at the start of the program, at 5 weeks and after 6 months.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parenting in Sweden (Experimental): The intervention group will be given the full program straight after recruitment ("Structured group discussions"). The program consists of five 3-hour sessions once a week. The themes for the five sessions are: Family in a new country, School, girls and boys, Health and health care system, Parents rights and obligations and parenting a teenager. Each session combines lectures and group discussions on topics critical to families adapting to life in Sweden. The sessions are held by a trained group leader and, if needed, interpreters.
  Interventions: Behavioral: Structured group discussions
- Waitlist (Placebo Comparator): The control group will be placed on a waiting list for 6 months ("Unstructured group meeting"). After 6 weeks the control group is offered a session with two short films from the Swedish Educational Broadcasting Company (UR), followed by a brief discussion. The first film explores how one can establish a place in society, the second film illustrates how hard it can be to create a new social context. The intention with the short films is not to give a short version of PiS, but to engage parents in the study and the program so they will complete them. The control group is then offered to participate in the whole program after 6 months.
  Interventions: Behavioral: Unstructured group meeting

INTERVENTIONS:
Behavioral: Structured group discussions — A group-based program for immigrant parents of children aged 0-17, providing essential information on key aspects of family life in Sweden. The intervention consists of five weekly three-hour sessions, combining lectures, group discussions, and interactive exercises, led by a trained group leader and, when necessary, an interpreter.
  The following topics are discussed:
  * Parenting in a New Country - Adapting to cultural changes and supporting children's integration.
  * Education & Child Development - School system, parental involvement, and learning support.
  * Healthcare & Well-being - Access to healthcare, preventive care, and mental health.
  * Parents' Rights & Responsibilities - Child welfare laws, positive discipline, and social services.
  * Parenting Teenagers - Navigating adolescence, peer relationships, and risk prevention.
  Other Names: Structured parenting support; Structured parenting guidance
  Arms: Parenting in Sweden
Behavioral: Unstructured group meeting — Parents in the control group are asked to participate in a gathering where they will watch two short films from the Swedish Educational Broadcasting Company (UR), followed by a brief discussion. The films have been handpicked by representatives from BRIS and PLUS together with the researchers to create an opportunity for a meeting. The first film "A way in - first meeting" shows a family from Iran living in Sweden for 1,5 years and explores how one can establish a place in society. In the second film "Make new friends" it is illustrated how hard it can be to create a new social context. The intention with the short films is not to give a short version of PiS, but to engage parents in the study and the program so they will complete them.
  Other Names: Community Orientation Session; Informational Meeting on Family Life in Sweden
  Arms: Waitlist

SUMMARY:
Supporting Parents in a New Country

Adjusting to parenthood in a new country presents significant challenges. Many immigrant parents face language barriers, financial difficulties, and cultural differences that can complicate their ability to support their children's adaptation to Swedish society. These challenges can contribute to increased stress within the family and, in some cases, elevate the risk of child maltreatment-particularly in socioeconomically disadvantaged areas. However, research suggests that strong social support and positive parenting strategies can mitigate these risks.

Sweden, known for its high levels of trust in authorities, has implemented various initiatives to assist families, especially those new to the country. One such initiative is Parenting in Sweden (PiS), a structured program designed to help foreign-born parents navigate Swedish society, understand their rights, and support their children's development. Delivered in five sessions, the program covers key topics such as the Swedish school system, healthcare services, parental rights, and challenges related to raising teenagers.

This study aims to assess whether participation in PiS increase parents' trust in social services. Additionally, it explores whether the program encourages parents to enroll their children in extracurricular activities, which are known to support child development. Another important aspect under investigation is whether the program can help reduce the risk of parents resorting to harsh disciplinary practices.

To evaluate these outcomes, the study follows a randomized controlled trial (RCT) design. Immigrant parents of children aged 0-17 are invited to participate, with half assigned to complete the full five-session program and the other half (control group) placed on a waiting list, receiving a group meeting to discuss films related to moving to Sweden. All participants will complete surveys assessing their trust in social services, their children's participation in extracurricular activities, and their parenting practices. These surveys will be administered before and after the program, as well as six months later, to track any changes over time.

The primary objective is to determine whether participation in PiS leads to increased trust in social services. Additional expected benefits (exploratory analysis) include promoting positive parenting behaviors, such as seeking help when needed and actively engaging children in structured activities outside of school.

By examining the effectiveness of parental support programs facilitating integration, this study aims to contribute to a deeper understanding of how structured interventions can help families navigate life in Sweden. If the program proves successful in fostering trust and encouraging positive parenting, it may have long-term benefits for both parents and children, ultimately supporting their well-being and integration into Swedish society.

ELIGIBILITY:
Inclusion Criteria:

* All parents invited to participate in PiS can take part in the study.
* Eligibility extends to parents born outside of Sweden who have children aged 0 to 17 years.
* There are no restrictions regarding the length of time since their migration to Sweden; i.e., participants may have lived in Sweden for decades prior to joining. - - Literacy is not a requirement for participation.

Exclusion Criteria:

* Individuals who are unable, physically or not willing, to sign a consent form will not be eligible to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
What are the effects of PiS on the level of trust in social services among parents born outside of Sweden? | From enrollment to 6 months after.
  The research question will be assessed through the question, "Overall, to what extent do you trust that those who work in Social services (SS) do their job?" ranked on a 5-point Likert scale.

SECONDARY OUTCOMES:
How valid and reliable is an adapted government trust scale for measuring trust in social services? | From enrollment to 6 months after.
  By using an adjusted version of a validated scale for the measure of trust in government, trust in social services will be assessed. The instrument measures on a 5-point Likert scale.
  English translation:
  * SS can help me feel well.
  * SS listen and try to understand what people say.
  * SS make decisions that help people.
  * SS is wise.
  * SS has sufficient knowledge to help me.
  * SS does their job well.
  * SS does what is best for people.
  * If people need help, SS does their best to help them.
  * SS makes decisions that help people manage on their own.
  * SS does everything to protect people.
  * SS cares about how people feel.
  * For SS, what politicians think is more important than how people feel.
  * SS tells it like it is.
  * SS does what they say they will do.
  * Those who work in SS are honest people.
  * It is possible to understand how SS has made their decisions.
Does participating in PiS increase enrollment of children in organized after-school activities | The question is asked in the baseline survey at enrollment and asked again at the 6-month follow-up.
  The number of children attending organized after-school activities will be measured through a forced-choice question: Do your children attend any organized after-school activities? If the answer is no, parents are given a number of options to tick .
Does participating in PiS decrease risk factors of child maltreatment? | From enrollment to 6 months after.
  Risk factors for use of child abuse will be assessed through a validated questionnaire, Brief Child Abuse Potential Inventory (BCAP) developed by Ondersma et al. BCAP is a shortened version of the screening tool for detecting potential child maltreatment, the Child Abuse Potential Inventory (CAPI). The CAP Inventory is a self-report measure of 160 forced-choice (agree/disagree) questions. But some characteristics, such as the length of the questionnaire and the complex scoring system, limit the screening tool's usefulness, which is why the shorter version was developed. BCAP contains seven factors: Distress, Family Conflict, Rigidity, Happiness, Feelings of Persecution, Loneliness, and Financial Insecurity. These factors are not used to produce individual factor scores but to ensure the Abuse Risk scale includes a range of dimensions associated with physical child abuse risk.

OTHER OUTCOMES:
What are the mechanisms behind the effectiveness of the program? | From enrollment to 6 months after.
  To understand the mechanisms behind the effectiveness of the program and to perform exploratory subgroup analysis, group leaders will also provide information. Through a baseline questionnaire, they are asked about their age, gender, which languages they speak, their native country and when they moved to Sweden if applicable, their highest education, their occupation, how many Parenting in Sweden groups they have led or if they have led any other groups in parental support programs, and how they assess their own knowledge regarding social services. They will also supply information through a self-assessment form regarding their leadership abilities, the content of the session, and parent engagement after every session.

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm - distibuted, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
Confidentiality. Sharing IPD would not align with ethical approval.